CLINICAL TRIAL: NCT03788746
Title: A Prospective, Non-Interventional Study to Assess the Prevalence of PD-L1 Expression in the First-Line Setting of Locally Advanced/Unresectable or Metastatic Urothelial Carcinoma
Brief Title: Prevalence of PD-L1 Expression in Patients With Advanced Urothelial Carcinoma
Acronym: PREVAIL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419BR00008
Record Dates: First submitted 2018-11-27; First posted 2018-12-28 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Carcinoma; Registry
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with advanced urothelial carcinoma: Patients with a confirmed diagnosis of advanced urothelial carcinoma, prior to or during first line therapy, who have available tumor tissue samples collected as part of standard of care

SUMMARY:
The purpose of this study is to assess the prevalence of pre-treatment tumor tissue PD-L1 expression in patients diagnosed with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
Advanced urothelial carcinoma (UC) (locally advanced/unresectable or metastatic UC) is a fatal disease with 5-year survival rate of 5%. The most frequently studied diagnostic for advanced UC is the programmed death-ligand 1 (PD-L1) protein expression in tumor tissue. A better understanding of PD-L1 expression in a "real world" setting could help understand its clinical utility in the management and decision making in advanced UC and clinical trial design

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Age ≥18 years old
* Patient must have advanced UC confirmed by their HCP; histologically- confirmed diagnosis of UC an dHCP-confirmed advanced UC.
* Patient must be either currently receiving 1L systemic treatment for their advanced UC or will be starting 1L systemic treatment (i.e. "newly diagnosed" advanced UC; 1L therapy is defined as the first systemic therapy given for advanced UC).
* Patient remains eligible for the study if they received neoadjuvant or adjuvant platinum-based chemotherapy if their recurrence was more than 12 months after their last chemotherapy dose.
* Radio-sensitizing chemotherapy as part of chemoradiation is NOT counted as neoadjuvant or adjuvant chemotherapy; thus, the 12-month interval mention above does not apply, and the patient would be eligible
* Patients with available tumor tissue sample (fresh or archival - up to 3 years old) that was collected as part of SoC any time prior to 1L treatment for advanced UC with a target of 18 slides (7 minimum) available for biomarker testing (PD-L1 and tTMB). Already prepared slides must have been cut within 6 months prior to PD-L1 testing.

Exclusion Criteria:

* Patients concurrently enrolled in other clinical trials that prohibit their participation in a non-interventional study
* Patient has resectable localized UC and has refused surgery
* Patients with history of non-urothelial active malignancy that completed therapy within 2 years from study enrollment except:

  * Any resected in situ carcinoma or non-melanoma skin cancer
  * Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy) and in which no systemic therapy was indicated

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population with care managed in a community setting in the United States
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Categorization of PD-L1 results (dichotomous, high vs. low) based on pre-treatment tissue samples. | 24 months
  The proportion of advanced UC patients with biomarker PD-L1 high results will be calculated.

SECONDARY OUTCOMES:
To assess the association of pre-treatment tumor tissue PD-L1 expression with pre-treatment tumor tissue TMB (tTMB) based on the chosen assay | 24 months
  Assay results for pre-treatment tTMB will be assessed by pre-treatment tumor tissue PD-L1 expression status.
To describe the objective response rate (ORR), progression-free survival (PFS) and overall survival (OS) as well as treatment patterns in the 1L setting of advanced UC | 54 months
  1L advanced UC treatment patterns (such as regimen/agents used, start (first dose) and stop (last dose) dates, reasons for cis/carboplatin ineligibility) will be collected.
  Objective Response: complete or partial response based on healthcare provider (HCP) assessment; Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria highly recommended Progression: evidence malignancy has become worse or spreads in the body (based on HCP assessment).
  Objective response and survival endpoints (overall, stratified by PD-L1 expression [high vs. low] including the following: ORR: The proportion of patients with a complete or partial response based on HCP assessment; PFS: The time from the start of 1L advanced UC treatment until progression or death (any cause); and OS: The time from start of 1L advanced UC treatment until death (any cause)
To assess the association between pre-treatment tumor tissue PD-L1 expression with objective response, PFS, and OS among treated patients (anti PD-L1/PD-1, chemotherapy, other) | 60 months
  Objective response, PFS, and OS (defined above) will be stratified by pre-treatment tumor tissue PD-L1 expression, and among patients treated with anti-PD-L1/PD-1 or chemotherapy or other.

OTHER OUTCOMES:
To assess the association of pre-treatment tumor tissue PD-L1 with pre-treatment bTMB | 24 months
  bTMB levels will be summarized among the subset of patients with blood available for testing using the chosen assay who are newly diagnosed with advanced UC and have yet to start 1L treatment. Results for TMB can range from 0 (non-shedder) to very high values >50 mut/Mb (no maximum has been determined). The results for pre-treatment bTMB will be presented by PD-L1 results (high vs low).
To assess changes in ctDNA levels (variant allele fractions [VAFs]) at 3 points of sample testing: (1) Before starting 1L treatment (pre-treatment) (2) before initiating treatment on day 1 of cycle 3, and (3) at the time of progression (if applicable) | 60 months
  ctDNA levels will be summarized among the subset of patients with blood available for testing using the chosen assay who are newly diagnosed with advanced UC and have yet to start 1L treatment. VAF is the relative frequency of alleles at a particular locus in a population, expressed as a percentage, ranging from 0.3% to 100%. Changes in ctDNA levels at 3 points of sample testing will be assessed.
To examine the correlation between pre-treatment tTMB and bTMB values | 24 months
  bTMB levels will be summarized among the subset of patients with blood available for testing using the chosen assay who are newly diagnosed with advanced UC and have yet to start 1L treatment. Assay results for pre-treatment tTMB will be assessed by pre-treatment bTMB results.
To assess the prognostic value of pre-treatment and changes to ctDNA levels, and pre-treatment tTMB compared to bTMB, for outcomes of ORR, PFS, and OS | 60 months
  bTMB and ctDNA levels will be summarized among the subset of patients with blood available for testing using the chosen assay who are newly diagnosed with advanced UC and have yet to start 1L treatment. Objective response, PFS, and OS (defined in secondary outcome measures) will be assessed by the following: changes to ctDNA levels (VAFs) at 3 timepoints (defined above); and pre-treatment tTMB assay results compared with pre-treatment bTMB assay results.

CONTACTS AND LOCATIONS:
Overall Officials: Petros Grivas, MD, Study Chair — University of Washington; Joshua Meeks, Study Chair — Northwestern University
Locations (57):
- United States (57):
  - Research Site, Little Rock, Arkansas
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Monterey, California
  - Research Site, Santa Rosa, California
  - Research Site, Denver, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Geneva, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Greenwood, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Brewer, Maine
  - Research Site, Lewiston, Maine
  - Research Site, Grand Rapids, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, East Brunswick, New Jersey
  - Research Site, Englewood, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Little Silver, New Jersey
  - Research Site, Mount Laurel, New Jersey
  - Research Site, Albany, New York
  - Research Site, Johnson City, New York
  - Research Site, Port Jefferson Station, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Temple, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BR00008&attachmentIdentifier=8334a74b-59dd-494b-add1-ab2a81e5a8a3&fileName=D3614C00003_(PXL_247606)-CSR_Synopsis_redacted_version_Final.pdf&versionIdentifier=